CLINICAL TRIAL: NCT03901300
Title: PLAY: An Intervention to Improve Motor Skills in Young Children
Brief Title: An Intervention to Improve Motor Skills in Young Children
Acronym: PLAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Amanda Staiano, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 2018-041; 1R21HD095035-01A1 (NIH)
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Physical Activity; Fundamental Motor Skills; Development, Child; Self-regulation
MeSH Terms: conditions — Motor Activity; Self-Control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fundamental Motor Skills (FMS) (Experimental): The FMS group will utilize the PLAY FMS app that provides instructional lessons, peer modeling videos, and activity breaks to deliver 720 minutes of targeted, structured FMS instruction time to the child over a 12 week period.
  Interventions: Behavioral: Fundamental Motor Skills App
- Unstructured Physical Activity (Active Comparator): The active comparator group will use a version of the PLAY app that provides instructional lessons to promote the equivalent dosage of unstructured physical activity for the child.
  Interventions: Behavioral: Unstructured Physical Activity App

INTERVENTIONS:
Behavioral: Fundamental Motor Skills App — Lessons will be provided over the app each week with notifications sent 5 days/week over 12 weeks specific to randomized experimental group.
  Arms: Fundamental Motor Skills (FMS)
Behavioral: Unstructured Physical Activity App — Lessons will be provided over the app each week with notifications sent 5 days/week over 12 weeks specific to randomized active comparator group.
  Arms: Unstructured Physical Activity

SUMMARY:
The goal of "PLAY" is to adapt and test a developmentally appropriate intervention delivered on a mobile app to parents, with the goal of teaching fundamental motor skill (FMS) proficiency to their preschool-aged children (ages 3 to 5 y). Seventy-two children (3 to 5 y of age) were randomized. Of these children, 36 parents were randomized to use the FMS app and 36 were randomized to use a version of the app that promotes unstructured PA as a comparator group. Parents in the FMS condition accessed instructional lessons, peer modeling videos, and activity breaks to deliver 720 minutes of targeted, structured FMS instruction time to their child over a 12-week period. Parents in the comparator arm used a version of the app that provides instructional lessons to promote the equivalent amount of unstructured PA for their child. Parents were asked to guide the intervention, as parental support, modeling, and co-participation predict children's engagement in PA.

DETAILED DESCRIPTION:
Preschoolers spend 4 hours/day in front of a screen, while fewer than one-quarter engage in the recommended two hours of daily physical activity (PA). The decline in PA, increase in screen-based behaviors, and onset of obesity during preschool years have been linked to lifetime risk of obesity and related comorbidities. However, emerging evidence indicates that "screen time" can actually be leveraged as a tool to increase children's PA and promote healthy weight. Specifically, PA interventions delivered over digital devices can provide real-time encouragement for children to be physically active. Prior interventions delivered over mobile devices were effective in increasing PA levels, including our own P-Mobile study that provided behavioral strategies to parents of children aged 6 to 10 years.

When considering how to support and motivate parents whose children are preschool-aged, teaching and modeling fundamental motor skills (FMS) are critical to enable children's PA. FMS like running, jumping, or throwing a ball, are basic, goal-directed movement patterns developed in early childhood that provide a foundation for children to be physically active and competent movers. These skills enable a child to function independently in their surrounding environment, engage with peers, and contribute to their ability to be physically active. Evidence has shown that children must establish a minimal level of FMS proficiency to continue participating in PA opportunities as they age. FMS and PA behaviors have a dynamic and reciprocal relationship. Children with higher levels of FMS are more physically active both during childhood and into adolescence. Therefore, a PA intervention for preschoolers should focus on developing FMS competence.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 years of age
* Physically capable of exercise
* Has no parent-reported mobility limitations that impairs performance of fundamental motor skills

Exclusion Criteria:

• Gross Motor Quotient at "gifted or very advanced" based on the Test of Gross Motor Development (TGMD-3)

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Staiano, PhD, Principal Investigator — Pennington Biomedical Study Director; E. Kipling Webster, PhD, Principal Investigator — Augusta University
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Webster EK, Kracht CL, Newton RL Jr, Beyl RA, Staiano AE. Intervention to Improve Preschool Children's Fundamental Motor Skills: Protocol for a Parent-Focused, Mobile App-Based Comparative Effectiveness Trial. JMIR Res Protoc. 2020 Oct 20;9(10):e19943. doi: 10.2196/19943. PMID 33079066
- [Result] Staiano AE, Newton RL, Beyl RA, Kracht CL, Hendrick CA, Viverito M, Webster EK. mHealth Intervention for Motor Skills: A Randomized Controlled Trial. Pediatrics. 2022 May 1;149(5):e2021053362. doi: 10.1542/peds.2021-053362. PMID 35415743
- [Result] Staiano AE, Saha S, Beyl RA, Kracht CL, Newton RL Jr, Webster EK. Parental engagement and implementation fidelity in a mHealth motor skills intervention for young children. Phys Educ Sport Pedagogy. 2025;30(4):390-402. doi: 10.1080/17408989.2023.2235394. Epub 2023 Jul 15. PMID 40777185

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A convenience sample was recruited using flyers at local childcare centers, email listserv, social media, and community health fairs.
Period: Overall Study
Arm/Group | Fundamental Motor Skills (FMS) | Unstructured Physical Activity
Started | 35 (Children were enrolled study participants. Parents were not study participants.) | 37
Completed | 32 | 37
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Only children were enrolled as study participants in the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fundamental Motor Skills (FMS) | Unstructured Physical Activity | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.8 (0.8) | 4.1 (0.8) | 4.0 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 33 | 36 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 21 | 24 | 45
  Race: African American | 8 | 11 | 19
  Race: Other | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 35 | 37 | 72
Fundamental Motor Skills (TGMD-3 Total Percentile Rank) [Mean (Standard Deviation); unit: percentile] — The percentile rank can vary from 1st to 99th percentile, with 1st indicating lowest motor skills and 99th indicating highest (best) motor skills.
  percentile | 18.6 (2.3) | 14.9 (2.1) | 16.7 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: App Adherence
Description: Adherence to the app intervention based on number of activity breaks completed over the 12 week intervention
Time Frame: From date of randomization until completion of the 12 weeks of intervention
Measure: Mean (Full Range); unit: percentage of activity breaks
Arm/Group | Fundamental Motor Skills (FMS) | Unstructured Physical Activity
Number analyzed (Participants) | 35 | 37
percentage of activity breaks | 71 [8 to 100] | 87 [8 to 100]

2. Secondary Outcome: Change in Test of Gross Motor Development (TGMD-3) Percentile Rank Between Baseline and Week 12
Description: A validated, reliable observation assessment to evaluate fundamental motor skills performance. Percentile ranks range from 1st (lowest) to 99th (highest/best).
Time Frame: baseline and 12 weeks (primary outcome)
Population: Delta in TGMD-3 Total Percentile Rank between baseline to Week 12
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Fundamental Motor Skills (FMS) | Unstructured Physical Activity
Number analyzed (Participants) | 32 | 36
percentile | 7.1 (1.4) | -5.5 (1.3)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Only the children were enrolled study participants, so AEs were only collected for the children.
Arm/Group | Fundamental Motor Skills (FMS) | Unstructured Physical Activity
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/37
Other Adverse Events (participants affected / at risk) | 0/35 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03901300/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03901300/ICF_001.pdf